CLINICAL TRIAL: NCT00787553
Title: Tinidazole Versus Cefazolin Antibiotic Prophylaxis of Vaginal and Abdominal Hysterectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Jose Antonio Simoes, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 920/2006
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Last update posted 2008-11-07 (Estimated); Status verified 2008-11

CONDITIONS: Hysterectomy
Keywords: hysterectomy; antibiotic prophylaxis; bacterial vaginosis; tinidazole; cefazolin
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Cefazolin; Tinidazole; Imidazoles

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- cefazolin (Active Comparator)
  Interventions: Drug: cefazolin
- tinidazole (Active Comparator)
  Interventions: Drug: tinidazole
- cefazolin plus tinidazole (Active Comparator)
  Interventions: Drug: cefazolin plus tinidazole

INTERVENTIONS:
Drug: cefazolin — 2.0 g, IV, 2 hours before surgery
  Arms: cefazolin
Drug: tinidazole — 2.0 g orally, 12 hours before surgery
  Other Names: imidazoles
  Arms: tinidazole
Drug: cefazolin plus tinidazole — cefazolin, 2.0 g IV 2 hours before surgery plus tinidazole 2.0 g orally 12 hours before surgery
  Other Names: cefazolin; tinidazole
  Arms: cefazolin plus tinidazole

SUMMARY:
Purpose: to compare the efficacy of tinidazole and cefazolin on the prophylaxis of the febrile and infectious morbidity after vaginal or abdominal hysterectomy. Methods: A randomized clinical trial carried out at the Women's Integrated Healthcare Center (CAISM)/UNICAMP, Campinas, Brazil. Women undergoing to total vaginal or abdominal hysterectomy were randomly enrolled into one of these three groups of antibiotic prophylaxis: tinidazole, cefazolin or an association of both.

DETAILED DESCRIPTION:
A randomized clinical trial carried out at the Women's Integrated Healthcare Center (CAISM)/UNICAMP, Campinas, Brazil, to compare the efficacy of tinidazole and cefazolin on the prophylaxis of the febrile and infectious morbidity after vaginal or abdominal hysterectomy. Women undergoing to total vaginal or abdominal hysterectomy were randomly enrolled into one of these three groups of antibiotic prophylaxis: tinidazole, cefazolin or an association of both.

ELIGIBILITY:
Inclusion Criteria:

* women undergoing to hysterectomy due to non-oncologic causes

Exclusion Criteria:

* previous pelvic infection
* antibiotic use within 7 days before surgery
* study drugs allergy
* immuno-incompetence
* urinary tract infection

Ages: 32 Years to 72 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2006-07; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Post-operative infection | one month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Simoes, MD, PhD, Principal Investigator — University of Campinas
Locations (1):
- University of Campinas, Campinas, São Paulo, Brazil